CLINICAL TRIAL: NCT04691024
Title: Effects of Remotely Applied Spinal Stabilization Exercises on Functional Level and Muscle Architecture in Individuals With Chronic Neck Pain
Brief Title: Remotely Spinal Stabilization Exercises in Individuals With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dilara Onan, Research Assistant, Physiotherapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-20111
Record Dates: First submitted 2020-12-22; First posted 2020-12-31 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Neck Pain
Keywords: neck pain; spinal stabilization exercises; tele-rehabilitation; muscle architecture; functional level
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Remotely Exercises 3 times a week, 8 weeks remotely (with video) spinal stabilization exercises
  Interventions: Other: Exercise
- Control Group (Other): Face to Face Exercises 3 times a week, 8 weeks face to face (in clinic) spinal stabilization exercises
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Spinal stabilization exercises

SUMMARY:
Neck pain is a problem that recurs at certain stages of life and can affect approximately half of the population. A problem in the cervical region can cause problems such as pain and limitation in the surrounding joints. Doing a job with functional activity or fulfilling professional requirements can aggravate neck pain. As a result, anatomical, physiological and psychological systems emerge as factors affecting pain. Determining the disability of the individual and the effectiveness of rehabilitation can be demonstrated with functional capacity assessment. It is stated that in individuals with chronic neck pain, architectural features such as functional cross-sectional area of deep neck muscles and reduction of muscle thickness change. Muscle preservation may increase as pain increases, and more protection too; Limitations can further increase conditions such as pain. In addition to the problem being only in the neck region, the whole spine posture may change, and the lumbar region muscles may also weaken by considering the spine as a whole. It is stated that the muscular architectural properties of the cervical and lumbar region, which play an important role in the posture of the spine in individuals with chronic neck pain, can be improved with exercise. During the 2020 years' pandemic process, the time spent at home, the use of mobile devices, the duration of working at home on a desk increased, and increases in spine pain reported to professionals were observed. The fact that family members are at home has increased the workload of the home and the frequency of performing functional activities has increased. It is reported that the distance between physiotherapists and patients should be at least 2 meters in clinics due to the risk of contamination. As a result, the pandemic process has brought the remote exercise management, tele-rehabilitation process to the fore for physiotherapists and the society. With spinal stabilization exercises, the functional level and muscle architecture of individuals with chronic neck pain can be associated with architectural changes in the spinal muscles. As a result of the 2020 years' pandemic, it is not known whether remote exercise and face-to-face exercises will have different effects on clinical variables, functional activities, muscle architecture, together with difficulties in accessing clinics. The aim of the study is to investigate the effects of remote spinal stabilization exercises on functional level and muscle architecture on individuals with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Having neck pain for at least 3 months,
* Between the ages of 18-55,
* Being literate,
* Individuals who are capable of understanding exercises (Montreal Cognitive Assessment Scale (MOCA) total score> 21) will be included in the study.

Exclusion Criteria:

* Cervical radiculopathy, thoracic outlet syndrome,
* Malignant condition,
* Having systemic diseases such as neurological, psychological, cardiovascular and loss of function due to these diseases,
* A history of surgery in the spine and upper extremity, including the cervical region, in the last 1 year period,
* Fracture in the spine and upper extremity, including the cervical region, with a history of inflammation,
* Acute infection,
* Continuing another rehabilitation program,
* Individuals who do not agree to participate in the study and do not give written consent will be excluded from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Evaluation of Muscle Thickness with Ultrasonography | 15 minutes, through study completion, an average of 8 weeks, Change from Baseline Muscle Thickness at 8 weeks
  Ultrasonography is used to evaluate the architectural properties of the muscle (such as thickness) in chronic painful musculoskeletal problems such as neck-back pain. Muscle architecture measurements with ultrasound will be carried out before and after the exercise program by the specialist radiology doctor who is blind to the results of the study using 3.5-10 MHz convex and linear probes (Soundcam Mobile Ultrasound Device). Within the scope of our study, the muscle thickness of the spinal muscles will be evaluated in the resting position.
Evaluation of the Functional Cross Sectional Area with Ultrasonography | 15 minutes, through study completion, an average of 8 weeks, Change from Baseline the FCSA at 8 weeks
  Ultrasonography is used to evaluate the architectural properties of the muscle (such as he Functional Cross Sectional Area (FCSA)) in chronic painful musculoskeletal problems such as neck-back pain. Muscle architecture measurements with ultrasound will be carried out before and after the exercise program by the specialist radiology doctor who is blind to the results of the study using 3.5-10 MHz convex and linear probes (Soundcam Mobile Ultrasound Device). Within the scope of our study, the muscle FCSA of the spinal muscles will be evaluated in the resting position.
Evaluation of Functional Capacity Level with Functional Capacity Assessment Test | 20 minutes, through study completion, an average of 8 weeks, Change from Baseline Functional Capacity Level at 8 weeks
  Functional capacity assessment evaluates the effectiveness (time to completion, weight it can handle) of each activity that includes different activities for neck pain. The test includes the activities of "repetitive reaching out, lifting objects overhead, working overhead". The validity and reliability of the Functional Capacity Assessment Test in individuals with chronic neck pain has been shown. The time individuals can complete the tests will be recorded.
Evaluation of Functional Capacity Level with Back Performance Scale | 10 minutes, through study completion, an average of 8 weeks, Change from Baseline Functional Capacity Level at 8 weeks
  The back performance test (Back Performance Scale) is a test that evaluates the effectiveness of each activity that includes 5 different activities (socks test, gathering test, righting test, fingertip-floor test, carrying test). The Back Performance Scale test is scored between 0-15 points. An increase in score indicates a poor result.

SECONDARY OUTCOMES:
Evaluation of pain severity | 5 minutes, through study completion, an average of 8 weeks, Change from Baseline pain severity at 8 weeks
  Pain Assessment: Visual Analogue Scale (VAS) VAS indicates the level of pain that the person is experiencing at the moment, marked with a vertical line on a plane. The pain felt by the person is marked as "0: I feel no pain", "10: I feel very severe pain". Scoring is based on measuring the participant's vertical marking for pain on the plane with a ruler. The validity and reliability study of the scale was conducted by Price et al.
Evaluation of disability | 5 minutes, through study completion, an average of 8 weeks, Change from Baseline disability at 8 weeks
  Disability Assessment: Neck Disability Questionnaire (NDI) Vernon et al. developed by. The Turkish version study was conducted by Aslan et al. Made by. The NDI includes a total of 10 questions such as pain, personal care, concentration, working, driving, sleeping. Each question is scored between 0-5 points. 0 points means no restrictions, 50 points means complete apology. 0-4 points are evaluated as no disability, 5-14 points as mild disability, 14-24 points as moderate disability, 25-34 serious disability and 35 and above as complete disability.
Evaluation of neck awareness | 5 minutes, through study completion, an average of 8 weeks, Change from Baseline neck awareness at 8 weeks
  Awareness Assessment: Fremantle Neck Awareness Questionnaire (FreNAQ) Likert type that evaluates the altered perception specific to the individual (0 = Never / I never feel like this, 1 = I rarely feel this way, 2 = Sometimes, or sometimes I feel this way, 3 = I often feel this way, 4 = I always or often feel this way) it is a survey. The questionnaire asks 9 questions to individuals such as how they perceive their neck according to their body, how they perceive their body position. The Fremantle Back Awareness Questionnaire, which is the original version of the questionnaire, was conducted by Wand et al. The Turkish validity and reliability of the neck version was developed by Onan et al.
Evaluation of quality of life | 5 minutes, through study completion, an average of 8 weeks, Change from Baseline quality of life at 8 weeks
  Quality of life Assessment: SF-36 SF-36 is a scale consisting of 36 questions that evaluates the health status of the person with 8 sub-items (physical function, role limitations, social function, mental health, vitality, pain, general health). Scoring between 0-100 is made separately for each sub-item. It indicates good health as the score approaches 100. The validity and reliability study, Koçyiğit et al. Made by.
Evaluation of Exercise Adherence Assessment: Exercise Adherence Rating Scale (EARS) (EUAS) | 5 minutes, through study completion, an average of 8 weeks, Change from Baseline Exercise Adaptation Assessment at 8 weeks
  It will be evaluated using the Exercise Adherence Rating Scale (EARS), which evaluates exercise compliance. The first 2 parts of the scale consist of 6 questions and the third part consists of 10 questions. The first part is not included in the scoring and the maximum score to be obtained from two parts is 64. An increase in score indicates an increased adaptation to exercise. The Turkish validity and reliability study of the scale was conducted in 2019 by Korkmaz et al.
Evaluation of Difficulty of Functional Activities and Exercise Program Satisfaction with Visual Analog Scale | 5 minutes, through study completion, an average of 8 weeks, Change from Baseline Difficulty of Functional Activities and Exercise Program Satisfaction at 8 weeks
  The Visual Analog Scale (VAS) is used in measurement by digitizing the values that cannot be measured numerically. It is a line measurement, often on a 10 cm long horizontal or vertical line, where the person indicates his condition. Pain is used in the literature to evaluate satisfaction. In the satisfaction evaluation, it is evaluated as "0: there was no decrease in complaints, I am not satisfied, 10: complaints completely disappeared, I am very satisfied". In the study, the functional activity difficulty will be evaluated as "0: Being unable to do the activity, 10: Being able to do the activity at the level before the neck pain started".
Evaluation of kinesiophobia | 5 minutes, through study completion, an average of 8 weeks, Change from Baseline kinesiophobia at 8 weeks
  Kinesophobia Assessment: Tampa Kinesophobia Scale (TCS) It is a 17-question scale that evaluates injury avoidance and fear of movement, and Kori et al. developed by. The Turkish version is from Tunca-Yılmaz et al. Made by. Its scoring is scored with "1 = Strongly disagree, 4 = Strongly agree". The score is calculated by reversing items 4, 8, 12 and 16. The total score is between 17 and 68. It is understood that the higher the score, the higher the kinesiophobia. A total score of more than 37 is considered to be a high degree of kinesophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Onan D, Ulger O, Martelletti P. Effects of spinal stabilization exercises delivered using telerehabilitation on outcomes in patients with chronic neck pain: a randomized controlled trial. Expert Rev Neurother. 2023 Mar;23(3):269-280. doi: 10.1080/14737175.2023.2192870. Epub 2023 Mar 22. PMID 36927237